CLINICAL TRIAL: NCT02866396
Title: Postoperative Oxycodone Consumption After Spinal Surgery in Pregabalin-treated Patients Compared to a 48-h Perioperative Administration: a Prospective, Observational Study
Brief Title: Impact of Pregabalin in Chronic Users vs. a Perioperative Limited Prescription on Oxycodone Requirement
Acronym: PREGAB
Status: Completed | Type: Observational
Sponsor: Christophe Aveline, MD (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor-Investigator, Christophe Aveline, MD, Principal investigator: Christophe Aveline, Department of anesthesia and surgical intensive care unit, Private Hospital, Private Hospital Sevigne
Organization: Private Hospital Sevigne (Other)
Other Study IDs: SPH-016-A
Record Dates: First submitted 2016-07-11; First posted 2016-08-15 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Pain; Neuropathic Pain
Keywords: chronic pain; oxycodone; pregabalin; lumbar spine surgery; multimodal analgesia
MeSH Terms: conditions — Pain, Postoperative; Neuralgia; Chronic Pain | interventions — Pregabalin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pregabalin patients: Same dose of preoperative pregabalin 1h after surgery associated to paracetamol 1g PO and ketoprofen 100mg PO Intraoperative: nefopam 20mg IV + ketamine 0.3mg/kg IV + dexamethasone 8mg IV Postoperative: morphine titration (PACU if NRS > 3) + paracetamol 1g/6h PO + ketoprofen 100mg/12h PO systematically, oxycodone 5-10mg/12h PO if NRS>3
  Interventions: Drug: Pregabalin
- Naive patients: Pregabalin 150mg PO initiated 1h before surgery and associated to paracetamol 1g PO and ketoprofen 100mg PO Intraoperative: nefopam 20mg IV + ketamine 0.3mg/kg IV + dexamethasone 8mg IV Postoperative: morphine titration in PACU (NRS > 3) + paracetamol 1g/6h PO + ketoprofen 100mg/12h PO systematically, oxycodone 5-10mg/12h PO if NRS>3
  Interventions: Other: Naive patient

INTERVENTIONS:
Drug: Pregabalin — Pregabalin continued at the same preoperative dose 1h before surgery associated to paracetamol 1g PO and ketoprofen 100mg PO Intraoperative: nefopam 20mg IV + ketamine 0.3mg/kg IV + dexamethasone 8mg IV Postoperative: morphine titration in PACU (NRS > 3) + paracetamol 1g/6h PO + ketoprofen 100mg/12h PO systematically, oxycodone 5-10mg/12h PO if NRS>3
  Other Names: ATC code: N03AX16
  Groups: Pregabalin patients
Other: Naive patient — Pregabalin 150mg PO initiated 1h before surgery Associated to paracetamol 1g PO and ketoprofen 100mg PO Intraoperative: nefopam 20mg IV + ketamine 0.3mg/kg IV + dexamethasone 8mg IV Postoperative: morphine titration in PACU (NRS > 3) + paracetamol 1g/6h PO + ketoprofen 100mg/12h PO systematically, oxycodone 5-10mg/12h PO if NRS>3
  Groups: Naive patients

SUMMARY:
Spinal surgery is associated with intense pain and associated to a history of preoperative chronic pain. Pregabalin is licensed to treat chronic neuropathic pain, particularly when high dose of opioid are required. Preoperative pain is associated with high postoperative pain scores and opioid requirement promoting persistent hyperalgesic state. The investigators will evaluate the postoperative opioid consumption and pain scores in patients scheduled for lumbar surgery and taking pregabalin since more than 15 days and compare with preoperative pregabalin-free patient that will receive pregabalin only during surgery.

DETAILED DESCRIPTION:
Patients will be prospectively included and compared according their preoperative medication: pregabalin-treated patients (>more than 15 days) for neuropathic pain associated to spinal surgery and pregabalin-free patients for whom pregabalin will be prescribed for 48 hours. Patients will be included without randomization as an observational study. All the patients will receive multimodal analgesia and intraoperative management will be standardized. The main outcome will be the amount of oxycodone during the first 24h after surgery. Other outcomes include pain scores, the quantification of the neuropathic pain diagnostic questionnaire (DN4), nausea and vomiting, length of stay, side-effects of pregabalin and opioid. Patients were also evaluated at three months for pain scores and DN4 score. Postoperative evaluation will be performed in a single-blind manner with investigators not include in the recruitment or the peroperative period.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiologist Physical status (ASA) 1-3
* Age ≥18 years old
* Spinal surgery: discectomy, posterior or transforaminal lumbar interbody fusion limited to 2 levels, lumbar disk prosthesis
* Able to participate personality, has given free and inform consent in French
* Affiliated of beneficiary of a system of social security

Exclusion Criteria:

* Age less than 18 years or higher than 85 years old
* Refusal to participate or provide written consent
* Surgery with a combined anterior and posterior approach
* Emergency surgery, reintervention, spine fracture, metastasis
* Tricyclic antidepressant use
* Pregabalin use for other indication: other neuropathy, epilepsy, generalized anxiety disorder
* Pregnancy
* Lack of understanding of NRS and/or DN4 scores
* Hypersensibility or contraindication to levobupivacaine, paracetamol, nefopam, ketoprofen and/or oxycodone
* Participation in another clinical study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will evaluate the postoperative opioid consumption and pain scores in patients scheduled for lumbar spine surgery and taking pregabalin since more than 15 days and compare with preoperative pregabalin-free patient that will receive pregabalin only during surgery.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Oxycodone consumption | 24h postoperatively
  mg

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) Pain at rest | the day before surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale (NRS) Pain during walking | the day before surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) at rest | 1h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) at rest | 4h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) at rest | 8h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) at rest | 12h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) at rest | 24h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) at rest | 48h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) at rest | 3 months after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) during walking | 12h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) during walking | 48h after surgery
  NRS: 0 no pain - 10 worst pain
Numeric Rating Scale Pain (NRS) during walking | 3 months ater surgery
  NRS: 0 no pain - 10 worst pain
remifentanil consumption | during surgery
  µg/kg/min
Morphine titration | 0-2h after surgery
  mg
Oxycodone requirement | 0-48h after surgery
  mg
Ondansetron requirement | 0-48h after surgery
  mg
DN4 score | preoperatively
DN4 score | on postoperative day one
DN4 score | on postoperative day two
DN4 score | three months after surgery
length of stay | on postoperative day five
  days
Post Opertive Nausea and vomiting (PONV) | 0-48h after surgery
  % of patients
Pregabalin side-effects | 0-48h after surgery
  diplopia, confusion, dizziness, psychiatric disorders (% of patients)
Sedation | 0-48h after surgery
  1: awake - 2: drowsiness, easily awake by appeal - 3: drowsiness, awake to tactile stimulation - 4: drowsiness, awake by pain

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Beloeil, MD, PhD, Study Chair — Rennes University Hospital; Christophe Aveline, MD, Principal Investigator — Private Hospital Sevigne
Locations (1):
- Christophe Aveline, MD, Cesson-Sévigné, France

IPD SHARING:
Plan to Share IPD: No